CLINICAL TRIAL: NCT06349239
Title: Maintenance Treatment With Oral Azacitidine for Patients With de Novo AML Including t-AML and AML-MRC in First Remission After CPX-351
Brief Title: Oral Azacitidine Maintenance Post-CPX 351
Acronym: ORAZ-351
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Hemato01
Record Dates: First submitted 2024-03-22; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: ONUREG; AML de novo
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Follow-up of disease

SUMMARY:
Approximately 10% of patient develop AML after chemotherapy or radiation for unrelated disease (t-AML) and 20% have AML with an antecedent hematologic disorder (AML-MRC). CPX-351 (Vyxeos), a liposomal formulation of a fixed molar ratio (1:5) daunorubicin and cytarabine, has been approved for treatment of adults with newly diagnosed t-AML or AML-MRC. CPX-351 significantly improved median overall survival.

Although induction chemotherapy results in remission in many older patients with AML, relapse is common and overall survival is poor. For patients not eligible for HSCT, maintenance therapies are needed to reduce the risk of relapse and prolong overall survival without causing undue adverse effects or compromising health-related quality of life. Oral azacitidine (ONUREG) has been approved by FDA on September, 2020, to treat adult patients with AML who achieved CR or CRi following intensive induction chemotherapy with or without consolidation and who are not able to complete intensive curative therapy (not candidate to HSCT).

The use of oral azacitidine maintenance is an integral part of clinical practice for AML patients who have achieved a first complete remission (CR) or complete remission with incomplete blood count recovery (CRi) after intensive ""3+7"" induction chemotherapy and who are unable to complete intensive curative therapy.

But there are few data on its efficacy as a post-CPX-351 maintenance agent in patients with newly diagnosed t-AML or AML-MRC or de novo AML.THe aim of this study is to show the improvement of overall survival with use of oral Azacitidine as maintenance for patients with de novo AML including t-AML or AML-MRC who achieved complete remission or complete remission with incomplete blood count recovery after CPX-351. Long-term product safety is also being studied

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > 64 years of age at the time of C1J1 CPX-351
* de novo AML including t-AML or AML-MRC according to WHO 2016
* Should have undergone induction therapy with CPX-351 with or without CPX-351 consolidation
* Patients in first line of treatment
* Should have achieved first CR/CRi/CRh status according to IWG criteria
* ECOG performance status of 0,1,2,3

Exclusion Criteria:

* Prior bone marrow or stem cell transplantation
* patients having achieved CR/CRi following an added therapy
* Patients alive at the start of the study who did not receive study information or who objected to the collection of data

Min Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with de novo AML, therapy-related AML or AML with myelodysplasia related changes in first remission (CR1, CRi1, CRh1 according to IWG) after CPX-351 induction with or without CPX-351 consolidation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | from first administration of ONUREG to death from any cause, assessed up to 60 moths
  evalute overal survival

SECONDARY OUTCOMES:
Safety and tolerance | from first administration of ONUREG to death from any cause, assessed up to 60 months
  number of patients with treatment related adverse events assessed by CTCAE v4.0 including clinical parameters and biological parameters

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No